CLINICAL TRIAL: NCT00000384
Title: Treatment of Pediatric Obsessive-Compulsive Disorder
Brief Title: Treatment of Obsessive-Compulsive Disorder (OCD) in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: R01MH055126 (NIH); R01MH055126 (NIH); R10MH055121 (NIH); DSIR 84-CTM
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2005-11

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Adolescence; Child; Cognitive Therapy; Combined Modality Therapy; Obsessive-Compulsive Disorder; Placebos; Sertraline; Patient Education; Psychotherapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy; Training Support; Sertraline

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy
Behavioral: Educational Support
Drug: Sertraline

SUMMARY:
The purpose of this study is to compare 3 treatments for children with OCD: medication (sertraline, SER) alone vs OCD-specific therapy (Cognitive Behavior Therapy, CBT) vs medication plus therapy. Some patients will receive an inactive placebo (PBO) instead of medication and/or Educational Support (ES, non-psychological treatment) instead of therapy.

One in 200 children suffer from OCD, but few receive appropriate treatment. Both CBT and medication seem to be effective, but their effectiveness, alone and in combination, has not been evaluated.

There are 2 phases to this trial. In Phase I the child will receive 1 of the following 6 treatments for 12 weeks: 1) SER alone; 2) pill PBO alone; 3) CBT alone; 4) SER plus CBT; 5) SER plus ES; 6) pill PBO plus ES. If the child responds to treatment, he/she will go on to Phase II in which the treatment will be slowly reduced, then stopped (discontinued), over time to test the treatment's durability. The child will be evaluated at Weeks 1, 4, 8, 12 (Phase I treatment), and Weeks 16, 20, 24, and 28 (Phase II discontinuation) to see how effective and durable the treatment is in treating your child's OCD.

A child may be eligible for this study if he/she:

Has obsessive-compulsive disorder (OCD) and is 8 - 16 years old.

DETAILED DESCRIPTION:
To contrast the degree and durability of improvement in pediatric obsessive-compulsive disorder (OCD), patients will be treated with 1 of 6 conditions (3 active treatments and 3 control treatments): sertraline alone (SER), OCD-specific Cognitive Behavior Therapy (CBT), both SER and CBT (SER plus CBT), pill placebo (PBO), pill PBO plus Educational Support (ES), and SER plus ES.

One in 200 youth suffers from OCD, yet relatively few receive appropriate treatment. Both CBT and medication appear beneficial in controlled studies; however, the relative efficacy of CBT and medication, alone and in combination (COMB) is unknown. Thus, well-designed treatment outcome studies are necessary to improve care for youth with OCD.

The experimental design covers 2 phases. Phase I is a 2 (site) x 2 (SER or pill PBO) x 3 (CBT, ES or non- psychosocial treatment) x 5 (repeated measures) factorial 12-week comparison of SER, CBT, COMB and the control conditions. In Phase II, responders advance to a 16-week discontinuation study to assess treatment durability. The primary outcome measure is the Yale-Brown Obsessive-Compulsive Scale. Assessments blind to treatment status take place at Week 0 (pretreatment); Weeks 1, 4, 8, 12 (Phase I treatment); and Weeks 16, 20, 24 and 28 (Phase II discontinuation). Besides addressing comparative efficacy and durability of the specified treatments, the investigators also examine time-action effects, differential effects on specific aspects of OCD, including functional impairment, and predictors of response to treatment.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must have:

DSM-IV diagnosed OCD.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1997-05; Study Completion 2002-04

CONTACTS AND LOCATIONS:
Overall Officials: Edna B. Foa, PhD, Principal Investigator; John S. March, MD, MPH, Principal Investigator
Locations (2):
- United States (2):
  - Duke Univ. Med. Ctr., Durham, North Carolina
  - Univ of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Garcia AM, Sapyta JJ, Moore PS, Freeman JB, Franklin ME, March JS, Foa EB. Predictors and moderators of treatment outcome in the Pediatric Obsessive Compulsive Treatment Study (POTS I). J Am Acad Child Adolesc Psychiatry. 2010 Oct;49(10):1024-33; quiz 1086. doi: 10.1016/j.jaac.2010.06.013. Epub 2010 Sep 6. PMID 20855047